CLINICAL TRIAL: NCT01935271
Title: Nutritional Supplementation and Muscle Health: A Pilot Study on Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 391351
Record Dates: First submitted 2013-02-20; First posted 2013-09-05 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Immunosenescence; Sarcopenia
Keywords: immunosenescence; sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Muscle Armor Supplement (Experimental): Treatment with a commercially available over the counter nutritional supplement
  Interventions: Dietary Supplement: Muscle Armor Supplement
- Placebo (Placebo Comparator): Sugar-based placebo drink mix
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Muscle Armor Supplement
  Arms: Muscle Armor Supplement
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The ability of older adults to improve their muscle strength through exercise training appears related to how well their immune system functions. Thus, a nutritional supplement which improves immune function could theoretically boost strength gained for older adults from exercise. The purpose of this pilot study is to determine if a nutritional supplement has any effect on immune function.

Veterans (age 60-80 yrs, N=12) be randomized in a double-blind placebo-controlled fashion to consume supplement or placebo for four weeks. After two weeks of consumption, subjects will be treated with a vaccine for tetanus, diphtheria, and pertussis. Blood will be drawn from each subject before and after vaccination to determine the effects of the supplement on immune response to vaccination. Additionally, subjects will undergo blood draw and muscle biopsy before and after two weeks of supplementation to determine the effects of supplementation on other measures of immune function (e.g. cytokine and growth factor levels). This is an important issue due to the serious health consequences associated with muscle loss in older adults and the need for improved strategies for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 60-80 years
* Body Mass Index of 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Participating in any other research study involving an intervention
* Smokes tobacco products
* Pains, tightness or pressure in chest during physical activity
* Participated in a weight-lifting targeting the thighs in last 3 months
* Problems walking or exercising with both legs
* Taking heparin, plavix / clopidogrel, or coumadin / warfarin
* Allergic to lidocaine
* Significant problem with fainting
* Allergic to vaccination
* Tetanus/diptheria/pertussis vaccine in previous two years
* Seizure in past 3 months
* Guillain-Barre Syndrome in past 3 months
* Enrolled in another interventional study
* Metastatic cancer or undergoing chemotherapy
* Cerebral aneurysm or intracranial bleed in past year
* End-stage congestive heart failure
* Unstable abdominal or thoracic aortic aneurysm
* Renal disease requiring dialysis
* Acute retinal hemorrhage or ophthalmologic surgery in past 3 months
* Bone fractures in the pelvis, legs, or feet in the last 3 months
* Hernia that causes pain during physical activity
* Myocardial infarction or cardiac surgery in past 3 months
* Pulmonary embolism or deep venous thrombosis in past 3 months
* Proliferative diabetic retinopathy or severe nonproliferative retinopathy
* Active suicidality or suicidal ideation
* Systemic bacterial infection
* Taking aspirin (in any form) and unable/unwilling to discontinue
* Unwilling to halt concurrent use of amino acid or protein supplements
* Unwilling to halt new use of nutritional supplements
* Unwilling to maintain current normal diet
* Encephalopathy in past 7 days
* Active oral or genital herpes
* Current use of appetite stimulants
* Current treatment for mania or bipolar disorder or taking lithium
* Diagnosis of a significant cognitive deficit
* Untreated severe aortic stenosis
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension or hypotension (>160/100, <100 systolic)
* Uncontrolled malignant cardiac arrhythmia
* Unstable angina (at rest or increased pattern in past month)
* Allergic to latex or tape
* Bleeding or clotting disorders
* Taking any nonsteroidal anti-inflammatories and unable to discontinue use
* Taking certain supplements and unable or unwilling to discontinue use
* Significant problems with chronic pain
* Uncontrolled asthma or allergies
* Taking lactulose, nitrates plus hypertension medications, or Viagra
* Liver cirrhosis or other severe liver disease
* History of peripheral artery disease
* Steroid or androgen use in past 3 months
* Other physician judgment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in antibody titer to tetanus, diptheria, pertussis antigen post-vaccination. | Baseline, 1 and 2 weeks post-vaccination
  The study will randomize subjects to consume supplement or placebo for 4-weeks. After two weeks of consumption, subjects will be vaccinated against tetanus, pertussis, and diphtheria. Blood will be drawn before and at two time points after vaccination. Change in antibody titer against the vaccine antigens will be calculated. A comparison between groups will determine if supplementation improves the antibody response to vaccination.

SECONDARY OUTCOMES:
Change in gene expression and protein levels in muscle and/or blood. | Baseline and after 2-weeks of supplementation
  The study will determine whether markers of inflammation in serum (e.g. C-reactive protein and cytokines) or blood mononuclear cells are decreased by the nutritional supplement. Blood will be drawn before and after periods of supplementation. The groups will be compared for protein and gene expression levels. The study will also determine whether supplementation affects muscle expression of genes associated with inflammation or tissue growth and remodeling. Muscle biopsies will be collected before and after two weeks of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dennis, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Dennis RA, Zhu H, Kortebein PM, Bush HM, Harvey JF, Sullivan DH, Peterson CA. Muscle expression of genes associated with inflammation, growth, and remodeling is strongly correlated in older adults with resistance training outcomes. Physiol Genomics. 2009 Jul 9;38(2):169-75. doi: 10.1152/physiolgenomics.00056.2009. Epub 2009 May 12. PMID 19435833